CLINICAL TRIAL: NCT02717234
Title: Appearance of Plasma Amino Acids Following Consumption of an Oral Nutrition Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 14.31.US.CLI
Record Dates: First submitted 2016-03-11; First posted 2016-03-23 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2016-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impact Advanced Recovery (Active Comparator): Oral nutrition supplement intended for consumption at 3 servings per day
  Interventions: Other: Oral Nutrition Supplement
- Impact Advanced Recovery-R (Experimental): Oral nutrition supplement intended for consumption at 3 servings per day
  Interventions: Other: Oral Nutrition Supplement

INTERVENTIONS:
Other: Oral Nutrition Supplement — Oral nutrition supplement intended for consumption at 3 servings per day

SUMMARY:
To assess the effect of consumption of an oral nutrition supplement on Arginine, a blood marker of nutritional intake

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject (absence of metabolic disorder, heart disease, endocrine disease, cancer)
* Discontinued use of omega 3 fatty acid supplements - 10 days prior to testing
* Willing to provide signed informed consent

Exclusion Criteria:

* Smoker
* Patients with potential for non-compliance
* Patients with allergy to ingredients in test products (i.e. milk protein, fish oil)
* Subject who in the Investigator's assessment cannot be expected to comply with study protocol
* Currently participating in another conflicting clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in plasma arginine levels in µmol/L | Pre-consumption, 30, 60, 120, 180, 240 minutes

SECONDARY OUTCOMES:
Change in plasma-free phospholipid Eicosapentaenoic acid (EPA) in µg/ml | Pre-consumption, 30, 60, 120, 180, 240 minutes
Change in plasma phospholipid Eicosapentaenoic acid (EPA) in µg/ml | Pre-consumption, 30, 60, 120, 180, 240 minutes

OTHER OUTCOMES:
Change in plasma-free phospholipid Docosahexaenoic acid (DHA) in µg/ml | Pre-consumption, 30, 60, 120, 180, 240 minutes
Change in plasma phospholipid Docosahexaenoic acid (DHA) in µg/ml | Pre-consumption, 30, 60, 120, 180, 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sherwyn Schwartz, MD, Principal Investigator — Diabetes & Glandular Disease Clinic, PA

IPD SHARING:
Plan to Share IPD: No